CLINICAL TRIAL: NCT02834689
Title: The Canadian E-PAraDiGM (Exercise Physical Activity and Diabetes Glucose Monitoring) Protocol
Acronym: E-PAraDiGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Alberta (Other); University of Calgary (Other); McMaster University (Other); Université de Sherbrooke (Other); Centre Hospitalier de l'Université Laval (Unknown); Children's Hospital Research Institute of Manitoba (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H1600377
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Walking; Seated Control
MeSH Terms: interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking (Experimental): Walking on a treadmill at 3.5 metabolic equivalents (METS) for 50 minutes
  Interventions: Behavioral: Walking
- Seated Control (Experimental): Sitting for 50 minutes
  Interventions: Behavioral: Seated Control

INTERVENTIONS:
Behavioral: Walking — Walking on a treadmill at 3.5 METS for 50 minutes
  Arms: Walking
Behavioral: Seated Control — Sitting for 50 minutes
  Arms: Seated Control

SUMMARY:
Walking is encouraged for people with type 2 diabetes but there is little evidence that performing a bout of walking can improve glucose control. Furthermore, it is unknown how participant characteristics (e.g., age, sex, medications) impact the acute glucose responses to walking in people with type 2 diabetes. The primary purpose of this study is to examine how a standardized bout of walking impacts glucose control assessed over 24 hours using continuous glucose monitoring. A secondary purpose is to determine whether responses are influenced by age, sex, and medication use.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with T2D for more than 6 months
* 30-90 years of age
* No contra-indications to exercise (PAR-Q+, Rose Angina questionnaire, limited ability to walk for 50 min).
* No previous myocardial infarction, stroke or diagnosed coronary artery disease
* No changes in diabetes medication in last 3 months
* Not treated by insulin or corticosteroids
* No significant change in body weight (>5%) in last 3 months
* Blood pressure <160/100 mmHg; resting HR<100
* Able to understand English or French and comply with study requirements (e.g., attend visits during the day)
* Hemoglobin A1C <9.0%
* No prior history of hypoglycaemia during activity or sleep

Exclusion Criteria:

* Chest pain during physical activity.
* Chest pain while resting (no physical activity) in the past month.
* Loss of balance or consciousness because of dizziness in past 12 months
* Bone or joint problem (for example, back, knee, or hip) that could be made worse by a change in physical activity.
* Currently pregnant or planning on becoming pregnant in the next 3 months
* Currently taking exogenous insulin
* Previous heart attack or stroke
* Any other reason that prevents ability to walk on a treadmill for 50 minutes

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Mean 24 hour glucose levels (mmol/l) | 24 hours
  Mean glucose assessed for 24 hours after walking or seated control assessed by continuous glucose monitoring

SECONDARY OUTCOMES:
Mean amplitude of glycemic excursions (MAGE) | 24 hours
  MAGE assessed for 24 hours after walking or seated control assessed by continuous glucose monitoring
Standard Deviation of Glucose Values | 24 hours
  Standard deviation of glucose values assessed for 24 hours after walking or seated control assessed by continuous glucose monitoring
Post-dinner glucose control | 2 hours following dinner
  Incremental area under the glucose curve for 2 hours following dinner
Post-lunch glucose control | 2 hours following lunch
  Incremental area under the glucose curve for 2 hours following lunch
Post-breakfast glucose control | 2 hour following breakfast
  Incremental area under the glucose curve for 2 hours following breakfast
Time spent above 10 mmol/l glucose | 24 hours following walking or seated control
  Time in minutes above 10 mmol/l assessed by continuous glucose monitoring over 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Rees JL, Chang CR, Francois ME, Marcotte-Chenard A, Fontvieille A, Klaprat ND, Dyck RA, Funk DR, Snydmiller G, Bastell K, Godkin FE, Dube MC, Riesco E, McGavock JM, Yardley JE, Sigal RJ, Gibala MJ, Weisnagel SJ, Prado CM, Jung M, Manders R, Lee T, Singer J, Boule NG, Little JP. Minimal effect of walking before dinner on glycemic responses in type 2 diabetes: outcomes from the multi-site E-PAraDiGM study. Acta Diabetol. 2019 Jul;56(7):755-765. doi: 10.1007/s00592-019-01358-x. Epub 2019 May 15. PMID 31093764